CLINICAL TRIAL: NCT02758665
Title: A Prospective, Open-label, Multicentre Phase-II Trial of Ibrutinib Plus Venetoclax Plus Obinutuzumab in Physically Fit or Unfit Patients With Previously Untreated Chronic Lymphocytic Leukemia (Cll) With tp53 Deletion (17p-) and/or Mutation
Brief Title: Trial of Ibrutinib Plus Venetoclax Plus Obinutuzumab in Patients With CLL
Acronym: CLL2-GiVe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: German CLL Study Group (Other); Roche Pharma AG (Industry); Janssen-Cilag Ltd. (Industry); AbbVie (Industry)
Responsible Party: Principal Investigator, Stephan Stilgenbauer, Prof. Dr. med., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2-GIVe
Record Dates: First submitted 2016-04-06; First posted 2016-05-02 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Leukemia, Lymphocytic, Chronic
Keywords: CLL; chronic lymphocytic leukemia; ibrutinib; venetoclax; obinutuzumab; TP53 Deletion
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obinutuzumab, Ibrutinib, Venetoclax (Experimental): Obinutuzumab i.v.: Cycle 1 (3000 mg), Cycle 2-6 (1000 mg) Ibrutinib (tablet): Cycle 1-15 (420 mg daily) Venetoclax (tablet): Cycle 1 (last 7 days 20 mg daily), Cycle 2 (ramp up 50 mg to 400 mg) Cycle 3-12 (400 mg daily)
  Interventions: Drug: ibrutinib; Drug: obinutuzumab; Drug: venetoclax

INTERVENTIONS:
Drug: ibrutinib
Drug: obinutuzumab
Drug: venetoclax

SUMMARY:
A prospective, open-label, multicentre phase-II trial of ibrutinib plus venetoclax plus obinutuzumab in physically fit (CIRS ≤ 6 & normal creatinine clearance) and unfit (CIRS > 6 & creatinine clearance ≥ 50 ml/min) patients with previously untreated chronic lymphocytic leukemia (CLL) with TP53 deletion (17p-) and/or mutation

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) with TP53 deletion (17p-) and/or mutation has a poor prognosis. Different therapeutic strategies have been tested over the last decade such as fludarabine-based regimens, alemtuzumab, bendamustine alone or with rituximab, lenalidomide, or ofatumumab, but all without compelling evidence for success. For example, with the FCR regimen as the standard 1st line treatment for fit CLL patients, only 5% (1 of 22) of patients with 17p deletion had a complete response (CR) and 40% of patients were free of disease progression at 12 months in the CLL8 Trial. New agents like Bruton's Tyrosin Kinase (BTK) inhibitors such as ibrutinib have shown promising results in patients with relapsed or refractory CLL, however, outcome of CLL patients with 17p deletion is inferior to other subgroups. The CLL11 trial revealed an impressive improvement in efficacy with GA-101 (obinutuzumab) as compared to rituximab when combined with Chlorambucil. Moreover, the BCL2 antagonist venetoclax (previously GDC-0199/ABT-199), tested as a single agent in relapsed / refractory CLL patients, showed striking activity with tumor lysis syndrome as dose limiting toxicity. Consequently, the current trial will test a combination regimen consisting of obinutuzumab, ibrutinib and venetoclax (the "GIVe" regimen) as first line treatment in CLL patients with TP53 deletion (17p-) and/or mutation with the aim to demonstrate efficacy in this population at highest unmet medical need.

The primary objective of the study is to evaluate the efficacy of the GIVe regimen in patients with TP53 deletion (17p-) and/or mutation and previously untreated CLL requiring treatment.

For this, the CR rate at cycle 15 (d1; final restaging) will be used as primary parameter for efficacy. The CR rate is defined as the proportion of patients having achieved a CR or a CR with incomplete recovery of the bone marrow (CRi) as best response (according to iwCLL criteria) until cycle 15 (d1; final restaging) from start of therapy.

Efficacy of the regimen will be further assessed by evaluation of the proportion of patients free of disease progression (PD-free rate) after 12 cycles of therapy, overall response rate (ORR), minimal residual disease (MRD) and overall survival as well as other time to event endpoints as outlined below.

A further secondary objective of the study is to evaluate the safety of ibrutinib, venetoclax and obinutuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Have documented CLL according to iwCLL criteria, measurable disease (lymphocytosis > 5x109 and/or palpable and measurable lymph nodes by physical exam and/or organomegaly assessed by physical exam)
2. Subjects must have untreated CLL, i.e. no prior chemotherapy, antibody therapy or non-chemotherapeutic agent (BTK, PI3K, BCL2 inhibitor or similar). Local irradiation or short term (up to 1 month) corticosteroid treatment for autoimmune phenomena are allowed
3. Subjects must have TP53 deletion (17p-) and/or mutation (in bone marrow or peripheral blood), with pre-existing local test results confirmed by central laboratory in Ulm
4. CLL requiring treatment ("active disease") according to the iwCLL criteria
5. ECOG ≤ 2
6. Creatinine clearance ≥ 50 ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured after 24 h urine collection
7. Adequate liver function as indicated by a total bilirubin ≤ 2 x, AST, and ALT ≤ 3 x the institutional ULN value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
8. No cardiovascular disability of New York Heart Association (NYHA) Class > 2. Class 2 is defined as comfortability at rest but moderate physical activity causes dyspnoea, angina pain or fatigue
9. Adequate bone marrow function (unless directly attributable to CLL, BM examination required):

   * ANC ≥ 1000/µl or
   * ANC < 1000/µl, if attributable to the underlying CLL (growth factor support may be administered after screening)
   * Platelets > 30.000/µl (unless directly attributable to the underlying CLL)
   * Hemoglobin ≥ 8g/dl (unless directly attributable to the underlying CLL)
10. Negative serological testing for hepatitis B (i.e. HBsAg negative and anti-HBc negative, patients positive for anti-HBc may be included if PCR for HBV DNA is negative) negative testing for hepatitis-C RNA and negative HIV test within 6 weeks prior to registration.

    [Patients who are HBsAg negative/anti-HBc positive with undetectable serum HBV DNA should be monitored closely (every month) for HBV DNA by a real-time PCR quantification assay with a lower limit of detection of the order of 10 WHO IU/mL until at least 24 months after the last treatment cycle with obinutuzumab. If the HBV DNA assay becomes positive, patients should pre-emptively be treated with a nucleoside analogue (i.e. lamivudine) for at 24 months after the last cycle of therapy with obinutuzumab or be referred to a gastroenterologist for management.]
11. Age at least 18 years
12. Life expectancy ≥ 6 months
13. Must be able to adhere to the study visit schedule and other protocol requirements
14. Able and willing to provide written informed consent and to comply with the study protocol procedures

Exclusion Criteria:

1. Transformation of CLL (i.e. Richter's transformation, prolymphocyctic leukemia)
2. One or more individual organ / system impairment score of 4 as assessed by the CIRS definition, excluding the Eyes, Ears, Nose, Throat and Larynx organ system
3. Known central nervous system (CNS) involvement
4. Patients with a history of PML
5. Active malignancies other than CLL within the past 2 years prior to study entry, with the exception:

   * Adequately treated in situ carcinoma of the cervix uteri
   * Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
   * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent and in remission at time of screening
6. Use of agents which would interfere with the study drug within 28 days prior to registration
7. Uncontrolled infection requiring systemic treatment
8. History of severe infusion-related reaction to humanized or murine monoclonal antibodies, and/ or known sensitivity or allergy to murine products or allergy to xanthin oxidase and rasburicase or glucose-6-phosphate dehydrogenase deficiency
9. Requires treatment with the following drugs:

   * Within 7 days prior to the first dose of study drug: No steroid therapy higher than 20 mg Prednisolone for anti-neoplastic intent; No CYP3A inhibitors (e.g. fluconazole, ketoconazole, clarithromycin, warfarin or phenprocoumon); No potent CYP3A inducers (e.g., rifampin, phenytoin or carbamazepine);
   * Within 3 days prior to the first dose of study drug: Grapefruit or grapefruit products; Seville oranges (including marmalade); Star fruit.
10. History of stroke or intracranial hemorrhage within 6 months prior to registration
11. Pregnant women and nursing mothers
12. Fertile men or women of childbearing potential unless:

    1. surgically sterile or ≥ 2 years after the onset of menopause
    2. willing to use two highly effective contraceptive methods (Pearl Index <1) during study treatment and for 18 months after end of study treatment.
13. Vaccination with a live vaccine a minimum of 28 days prior to registration
14. Legal incapacity
15. Prisoners or subjects who are institutionalized by regulatory or court order
16. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate | at day 1 of cycle 15 (1 cycle = 28 days) after start of induction therapy

SECONDARY OUTCOMES:
PD-free rate | up to 336 days
  Proportion of patients free of disease progression (PD-free rate) after 12 cycles of therapy
Overall Response rate | up to 1176 days
  Overall response rate (ORR) (including all patients achieving a complete response (CR), a complete response with incomplete recovery of the bone marrow (CRi), a partial response (PR) and a PR with lymphocytosis)
ORR | at 1008 days (=end of maintenance treatment)
  ORR after end of maintenance treatment
MRD levels | at the following days: 252, 336, 393, 381 as well as in bone marrow at day 393
  MRD levels (measured in peripheral blood after cycle 9, after cycle 12, at the beginning of cycle 15 (d1), at the beginning of cycle 36 (d1), as well as in bone marrow at the beginning of cycle 15)
Progression-free survival (PFS) | up to 1176 days
  Progression-free survival (PFS)
Event-free survival (EFS) | up to 1176 days
  Event-free survival (EFS)
Overall survival (OS) | up to 1176 days
  Overall survival (OS)
Duration of response in patients with (clinical) CR/CRi, PR | up to 1176 days
  Duration of response in patients with (clinical) CR/CRi, PR
Time to next CLL treatment (TTNT) | up to 1176 days
  Time to next CLL treatment (TTNT)
Treatment-free survival (TFS) | up to 1176 days
  Treatment-free survival (TFS)
Subsequent Treatment for CLL | up to 1176 days
  Evaluation of subsequent treatment for CLL (including proportion receiving allogeneic SCT as consolidation or in relapse) including response to treatment
Safety Parameters (Type, frequency, and severity of adverse events (AEs) and adverse events of special interest (AESI) and their relationship to study Treatment) | up to 1176 days
Incidence of Richter's transformation | up to 1176 days
  Incidence of Richter's transformation

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (11):
  - Universitätsklinikum Köln, Cologne
  - BAG Onkologische Gemeinschaftspraxis, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg / Saar
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum Schwabing, München
  - Unimedizin Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092